CLINICAL TRIAL: NCT04402034
Title: Telerehabilitation in Disabled People: Proposal for Practical Intervention With Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carlos Bandeira de Mello Monteiro, Associate Professor, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03851012.7.0000.5390
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Disability Physical
Keywords: Disability Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Application of tele-rehabilitation (Experimental): Individuals that will perform the protocol of virtual reality intervention.
  Interventions: Behavioral: Application of tele-rehabilitation

INTERVENTIONS:
Behavioral: Application of tele-rehabilitation — Individuals that will perform the virtual reality intervention.

SUMMARY:
This is a cross-sectional study, that is going to be conducted during the quarantine, period established by the state of São Paulo to reduce the transmission of COVID-19, between March 24 2020 and May 31 2020. Thus, the differential of this study is to use 100% telerehabilitation, in which the rehabilitation team and participants only had telephone contact, communication application (WhatsApp) and software interaction. 40 participants will be included. Potential and interested volunteers will be assessed by a detailed screening using the eligibility criteria and attended an initial selection for enrolment in the study. It wiil be used a platform called MoveHero, available for free use in https://movehero.com.br/. The individual needs access the internet, and once he gets online, he had to create his own account, inserting his name, email and creating a password. Considering that the platform presents different levels of difficulty, after the participant is connected to the platform, the researcher directed the participant to the protocol bespoke for each participant, playing 3 rounds of the game for 5 minutes each (total of 15 minutes). During the intervention, it will be applied BORG scale in order to assess their perceived effort.

DETAILED DESCRIPTION:
Instrument In this study, it will be used a platform called MoveHero, available for free use in https://movehero.com.br/. The individual needs access the internet, and once he gets online, he had to create his own account, inserting his name, email and creating a password. Considering that the platform presents different levels of difficulty, after the participant is connected to the platform, the researcher directed the participant to the protocol specially developed for cerebral palsy. MoveHero is considerate a timing coincident task and present several spheres falling down on the computer screen, with a musical rhythm to increase engagement. Thus, the participants will be positioned in front of a computer and when the game started the webcam captures the participant movements and a representation of the players appears on the computer screen as an avatar. The game goals are to intercept all falling spheres using upper limb wave movements in the exact moment the spheres reached their specific target in the bottom of computer screen. The game presented four columns with fixed targets in parallel allocated in two height levels (e.g. two on the left - targets A and B; two on the right - targets C and D). The game provides hit and miss feedback - if the individual reaches the spheres correctly, the game presented a feedback with the spheres changing the color for green (hit information). On the other hand, if the participant do not touch the spheres properly, the spheres changing the color for red and the letter X appears inside the target (miss information).

Software score During the game match (each game match lasts for 5 minutes) the participant can follow the score determined by the number of spheres hit (i.e. the information from each sphere hit appears in the bottom left side of the screen all the time) and at the end of each game match the participant had feedback with their total score (when the game match finished a total score appears in the middle of the computer screen). The game features 10 different and progressive phases of difficulty, considering the number of balls falling. In this study, all participants will start at the easiest phase (phase 1) and according to their own score, the researcher should move forward to a more difficult phase. The progression in the phase was established by the table below. Thus, each participant presents an individual progression, considering their performance.

Assessments

To characterize the participants it will be used some scales that characterize each disease and can be applied such as Pediatric Evaluation of Disability Inventory (PEDI) for children and Quality of Life and specific scales for adults. As well as sociodemographic Information: some questions will be asked, such as age, sex, income to understand the studied population.

To analyse the outcome Measures will be used: 1) Brunel Mood Scale (BRUMS) measures six identifiable affective states (Tension, Depression, Anger, Vigor, Fatigue, and Confusion) through a 24-item self-report inventory, with respondents rating a list of adjectives on a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely), based on subjective feelings. The instructions refer to how participants have been feeling in the past week, including today. 2) BORG scale: is Rating of Perceived Exertion used to measure the subjective intensity of effort. It is based on the sensations felt during exercise, such as muscle fatigue, increased heart rate and increased breathing. 3) System Usability Scale (SUS), was proposed by John Brooke in 1986 as the usability test tool. It is a simple scale based on a questionnaire and has been widely adopted in product usability evaluations. The statements cover a variety of aspects of system usability such as the need for support, training, and complexity, and thus have a high level of face validity for measuring usability of a system. The SUS instrument is generally used after the respondent has had an opportunity to use the system being evaluated. This instrument is a highly robust and versatile tool for usability professionals.

1.5 Procedure and Design

Contact and assessment scales

The parent's individuals (for children) or the individual itself will be contacted by phone and asked to perform the task at home, they will be assisted by the researcher over the phone, with a video call. Important to emphasized that all participants that need assistance, will be assisted by their parents or their caregivers. First, they wiil receive a link with research information and the assent and consent form to fill out and the inclusion criteria will be checked by researcher. When they agree to participate, a link to access a questioner will be sent with Brunel Mood Scale, BORG scale, PEDI and Sociodemographic Information. When parents and participants finish those scales the gaming platform will be accessed and the participant starts the protocol practice.

Practicing the task

Participants will perform the task individually in their own house with a family member helping and giving support during all protocol. The researcher contacts the family member and gives the following instructions using videocall (research interact with the family member and the participant during all the protocol): 1) place the computer on a table and login to the platform; 2) position the cell phone (to provide videocall) on the side of the computer to receive instructions; 3) provide a comfortable sitting position in a chair (individual should be positioned at a distance of approximately 1.5 m meters from the computer monitor) and adjusted in height according to the needs of the individual (if applicable, participants could use their own wheelchair); 4) after being seated and connected to the platform the research will explain the task verbally for all participants and ask the family member to play ones (demonstrations of how to perform the coincidence timing was given form the family member during two minutes); 5) after demonstration, the family member should grab the mobile phone (to have the opportunity to move the phone and show the participant performance to the researcher during all the protocol) and 6) thus, the therapist (by video call) instructed the participant to stay still and wait the first sphere appears on the screen. Once the first sphere appears, the individual had to move his or her hand to either touch the sphere exactly at the moment coinciding with the bottom target and the game should move on with different spheres falling in the computer screen.

Protocol

As presented before the parent and participant should answer 4 assessments (Brunel Mood Scale, BORG scale, PEDI and Demographic Information), and start to perform the first game phase (phase 1), after 5 minutes playing the game the participant will answer the Borg scale and researcher will analyze the game score (e.g. according to table 2 the participant should repeat phase one or move forward for a more difficult phase); the participant started a second practice and after 5 minutes answer the Borg scale (again- the participant should repeat last phase or move forward for a more difficult phase); the participant started a third and last practice and after 5 minutes had to answer the Borg scale and to finish the protocol the BRUMS scale and the System Usability Scale (SUS).

ELIGIBILITY:
Inclusion Criteria:

* agreement to participate
* clinical diagnosis of the disease
* age ranging from 7 to 80 years old

Exclusion Criteria:

* do not understand the tasks
* motor difficulties that impede the completing of the virtual tasks
* do not have technology devices to perform the virtual task (computer) or to contact the researcher (cell phone or a second computer)
* was precluded from completing the task due to some technological failure (such as internet crash).

Ages: 7 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Motor performance. | 1 day
  The motor performance will be measured by the virtual game "MoveHero", which gives data about accuracy, precision and directional trend of movement.

SECONDARY OUTCOMES:
Perceived Exertion. | 1 day.
  The Perceived Exertion will me assessed by the Borg Rating of Perceived Exertion (RPE), based on a 6 to 20 rating scale, in which a rating of 6 perceiving "no exertion at all" to 20 perceiving a "maximal exertion" of effort.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos BM Monteiro, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Escola de Artes,Ciencias e Humanidades da Universidade d Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] da Silva TD, da Silva PL, Valenzuela EJ, Dias ED, Simcsik AO, de Carvalho MG, Fontes AMGG, Alberissi CAO, de Araujo LV, Brandao MVDC, Dawes H, Monteiro CBM. Serious Game Platform as a Possibility for Home-Based Telerehabilitation for Individuals With Cerebral Palsy During COVID-19 Quarantine - A Cross-Sectional Pilot Study. Front Psychol. 2021 Feb 2;12:622678. doi: 10.3389/fpsyg.2021.622678. eCollection 2021. PMID 33633648